CLINICAL TRIAL: NCT03621215
Title: The Effect of Tart Cherry Juice on Risk of Gout Attacks: a Randomised Controlled Trial
Brief Title: The Effect of Tart Cherry Juice on Risk of Gout Attacks
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to COVID restrictions
Sponsor: Sheffield Hallam University (Other)
Collaborators: Cherry Research Committee (Other)
Responsible Party: Principal Investigator, Tony Lynn, Principal Lecturer (Food and Nutrition Group), Sheffield Hallam University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ER7166682; AA4736173 (Other Grant/Funding Number: Cherry Research Committee/Cherry Marketing Institute)
Record Dates: First submitted 2018-07-30; First posted 2018-08-08 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Gout Flare; Gout Attack
Keywords: tart cherries; gout; cardiovascular disease risk; gout attack; gout flare
MeSH Terms: conditions — Gout

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to consume either tart cherry juice or a fruit-flavoured placebo drink (matched as closely as possible for energy and sensory characteristics) daily for 12 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tart cherry juice (Experimental): 30 mL tart cherry concentrate (CherryActive, UK) diluted with 220 mL of water once per day (250 mL total volume per day). According to available manufacturers data, this is equivalent to consuming 90-100 fresh cherries per day.
  Interventions: Dietary Supplement: Tart cherry juice
- Fruit-flavoured placebo drink (Placebo Comparator): Matched for sensory characteristics and energy (with the addition of glucose).
  once per day (250 mL total volume per day)
  Interventions: Other: Fruit-flavoured placebo drink

INTERVENTIONS:
Dietary Supplement: Tart cherry juice — 30 mL tart cherry juice concentrate (CherryActive, UK), diluted with water to 250 mL. This is consumed daily by participants, with breakfast, for 12 months.
  Arms: Tart cherry juice
Other: Fruit-flavoured placebo drink — Consumed daily by participants, with breakfast, for 12 months.
  Arms: Fruit-flavoured placebo drink

SUMMARY:
The purpose of this study is to determine whether consuming tart cherry juice daily for 12 months reduces the risk of gout attacks during this period. Individuals with an existing gout diagnosis and who have experienced at least one gout flare in the past year will be recruited to participate in this study.

DETAILED DESCRIPTION:
Gout is a painful and often debilitating condition affecting around 3% of adults in the UK. It is a type of inflammatory arthritis caused by high levels of uric acid which is deposited as crystals in joints, resulting in painful gout flares. Cherries and cherry products have received attention for their possible role in gout management owing to their anti-inflammatory and anti-oxidant properties. Their consumption has been associated with a lower risk of gout attacks in one observational study. The consumption of cherries is also endorsed by several gout information websites and in the British Society of Rheumatology's 2017 guidelines for the management of gout. However, there is limited evidence underpinning these claims and existing studies tend to be short in duration and have small participant numbers. Gout attacks are sporadic in nature and so a long-term trial is required to clarify the therapeutic effect of cherries on gout attack risk.

The investigators are aiming to recruit 120 participants who have had at least one gout flare in the previous 12 months. Using the work of Rothenbacher et al., 2011, the chance of these individuals experiencing at least one attack in the next 12 months has been calculated at 11%. It is predicted that treatment with daily cherry juice consumption will reduce gout flare recurrence (primary outcome measure) to 1/4 of the rate of the actual recurrence i.e. to 2.7%. Using these figures, a sample size of 93 participants would provide power of 0.95 at a significance level of 0.05. A sample size of 120 participants allows for an approximate 20% attrition rate.

Participants will consume either 30 mL tart cherry juice (CherryActive) diluted to 250 mL with water or a fruit-flavoured placebo drink daily with breakfast for 12 months. Participants will be followed up at 6 and 12 months at the investigators' laboratory to study changes in gout flare frequency and intensity, uric acid levels and levels of inflammation. This will help determine if tart cherry juice could help reduce or even prevent gout attacks. Additionally, as gout is associated with increased cardiovascular disease (CVD) risk, changes in CVD risk markers, including blood pressure, arterial stiffness and cholesterol levels, will also be assessed.

Participants will be recruited through the use of posters, advertising on the UK Gout Society website, emails to large organisations and through letters sent from General Practitioners' (GP) surgeries to eligible patients. Potentially eligible patients will be identified by surgery staff using their patient database before contact information is passed to the research team at the surgery to prepare and send out invitation letters. As this method of recruitment involves accessing patient identifiable data (name and home address) prior to patient consent being given, an application to the Confidentiality Advisory Group (CAG) will be submitted for consideration.

A general linear mixed model analysis will be used to assess the effect of treatment allocation, time and their interaction on both primary and secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* existing diagnosis of gout
* have experienced at least one gout flare in the previous 12 months
* able and willing to participate in the study and provide written informed consent

Exclusion Criteria:

* frequently consume cherries or cherry products e.g. cherry supplements and juice (more than once a week)
* severe renal impairment (estimated glomerular filtration rate of <30ml/min)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
Change in gout flare frequency | Measured at 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 months
  Difference in gout flare frequency in tart cherry juice group versus placebo group from baseline to 12 months. Recorded as number per month.

SECONDARY OUTCOMES:
Change in gout flare intensity | Measured at 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 months
  Difference in gout flare intensity in tart cherry juice group versus placebo group from baseline to 12 months. Using a 0-10 Likert pain scale. The scale measures the pain of any gout flare. The possible score ranges from 0 for no pain through to 10 for worst pain imaginable. Change in pain scores between treatment and placebo groups will be compared throughout the duration of the intervention.
Changes in serum urate (in millimoles per litre (mmol/l)) | Measured at 0, 6 and 12 months
  Difference in serum urate in tart cherry juice group versus placebo group from baseline to 12 months.
Change in fractional excretion of uric acid (as a percentage, %) | Measured at 0, 6 and 12 months
  Difference in fractional excretion of uric acid in tart cherry juice group versus placebo group from baseline to 12 months. Measured from 24 hour urine sample.
Change in inflammatory markers (in milligrams per litre (mg/l)) | Measured at 0, 6 and 12 months
  Difference in inflammatory markers (c reactive protein (CRP), inter leukin-6 (IL-6) and tumour necrosis factor- alpha (TNF-alpha)) in tart cherry juice group versus placebo group from baseline to 12 months. Measured using an enzyme-linked immunosorbent assay (ELISA).
Change in oxidative damage (in percentage (%) of tail DNA) | Measured at 0, 6 and 12 months
  Difference in markers of oxidative stress in tart cherry juice group versus placebo group from baseline to 12 months. Measured using single-cell electrophoresis 'comet assay' as 8-oxo-dg levels in lymphocytes.
Change in antioxidant status (in percentage (%) of tail DNA) | Measured at 0, 6 and 12 months
  Difference in antioxidant status in tart cherry juice group versus placebo group from baseline to 12 months. Measured using single-cell electrophoresis 'comet assay' as resistance of DNA lymphocyte to H202-induced DNA strand breaks.
Change in blood pressure (in millimetres of mercury (mmHg)) | Measured at 0, 6 and 12 months
  Difference in brachial and central blood pressure in tart cherry juice group versus placebo group from baseline to 12 months. Measured using a Vicorder.
Change in arterial stiffness (in meters per second (m/s)) | Measured at 0, 6 and 12 months
  Difference in arterial stiffness in tart cherry juice group versus placebo group from baseline to 12 months.
Change in lipid profile (in millimoles per litre (mmol/l)) | Measured at 0, 6 and 12 months
  Difference in total cholesterol, HDL cholesterol, LDL cholesterol and triacylglycerides) in tart cherry juice group versus placebo group from baseline to 12 months.
Height (in meters (m)) | Measured at 0, 6 and 12 months
  Height and weight will be combined to report BMI in kg/m^2. Difference in BMI in tart cherry juice group versus placebo group from baseline to 12 months.
Weight (in kilograms (kg)) | Measured at 0, 6 and 12 months
  Height and weight will be combined to report BMI in kg/m^2. Difference in BMI in tart cherry juice group versus placebo group from baseline to 12 months.

OTHER OUTCOMES:
Changes in habitual diet | Measured at 0, 6 and 12 months
  4 day diet diaries will be used to assess any changes in habitual diet as a result of, or over the course of, the study.
Changes in habitual physical activity levels | Measured at 0, 6 and 12 months
  4 day physical activity logs will be used to assess any changes in habitual activity levels as a result of, or over the course of, the study.

CONTACTS AND LOCATIONS:
Overall Officials: Margo Barker, Principal Investigator — Sheffield Hallam University
Locations (1):
- Food and Nutrition Group, Sheffield Hallam University, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Neogi T, Chen C, Chaisson C, Hunter DJ, Choi HK. Cherry consumption and decreased risk of recurrent gout attacks. Arthritis Rheum. 2012 Dec;64(12):4004-11. doi: 10.1002/art.34677. PMID 23023818
- [Background] Jacob RA, Spinozzi GM, Simon VA, Kelley DS, Prior RL, Hess-Pierce B, Kader AA. Consumption of cherries lowers plasma urate in healthy women. J Nutr. 2003 Jun;133(6):1826-9. doi: 10.1093/jn/133.6.1826. PMID 12771324
- [Background] Kuo CF, Grainge MJ, Mallen C, Zhang W, Doherty M. Rising burden of gout in the UK but continuing suboptimal management: a nationwide population study. Ann Rheum Dis. 2015 Apr;74(4):661-7. doi: 10.1136/annrheumdis-2013-204463. Epub 2014 Jan 15. PMID 24431399
- [Background] Cea Soriano L, Rothenbacher D, Choi HK, Garcia Rodriguez LA. Contemporary epidemiology of gout in the UK general population. Arthritis Res Ther. 2011 Mar 3;13(2):R39. doi: 10.1186/ar3272. PMID 21371293
- [Background] Rothenbacher D, Primatesta P, Ferreira A, Cea-Soriano L, Rodriguez LA. Frequency and risk factors of gout flares in a large population-based cohort of incident gout. Rheumatology (Oxford). 2011 May;50(5):973-81. doi: 10.1093/rheumatology/keq363. Epub 2011 Jan 12. PMID 21228059
- [Background] Dalbeth N, Ames R, Gamble GD, Horne A, Wong S, Kuhn-Sherlock B, MacGibbon A, McQueen FM, Reid IR, Palmano K. Effects of skim milk powder enriched with glycomacropeptide and G600 milk fat extract on frequency of gout flares: a proof-of-concept randomised controlled trial. Ann Rheum Dis. 2012 Jun;71(6):929-34. doi: 10.1136/annrheumdis-2011-200156. Epub 2012 Jan 23. PMID 22275296
- [Derived] Lamb KL, Lynn A, Russell J, Barker ME. Effect of tart cherry juice on risk of gout attacks: protocol for a randomised controlled trial. BMJ Open. 2020 Mar 15;10(3):e035108. doi: 10.1136/bmjopen-2019-035108. PMID 32179562